CLINICAL TRIAL: NCT05528068
Title: Effect of Lifestyle Intervention Based on Continuous Physiological Monitoring Among Patients With Hypertension or High-normal Blood Pressure
Brief Title: Effect of Lifestyle Intervention Among Patients With Hypertension or High-normal Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Xue Feng, Executive Deputy Director, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-1559
Record Dates: First submitted 2022-08-25; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Hypertension; High-normal Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): standard care, physiological monitoring by wearable devices and healthy lifestyle education
  Interventions: Behavioral: healthy lifestyle education
- supervised lifestyle intervention group (Experimental): standard care, physiological monitoring by wearable devices and personalized and supervised lifestyle intervention including dietary and physical activity modification
  Interventions: Behavioral: supervised lifestyle intervention

INTERVENTIONS:
Behavioral: supervised lifestyle intervention — Participants will receive personalized dietary and exercise prescription according to the assessment of nutritional status, physical fitness and physiological-biochemical indexes. The participants will use the digital application for the first 3 months with supervised lifestyle intervention. Wearable devices, such as ambulatory blood pressure monitoring, dynamic electrocardio scanner and smart watch, will be worn to provide continuous physiological monitoring for safety. And then, participants will use the application by self-management for the next 6 months. All participants are given questionnaires, nutritional, physical fitness and physiological-biochemical assessment at baseline, 3 months, 6 months and 9 months.
  Arms: supervised lifestyle intervention group
Behavioral: healthy lifestyle education — Participants will receive standard care and healthy lifestyle education for hypertension prevention and control. Wearable devices, such as ambulatory blood pressure monitoring, dynamic electrocardio scanner and smart watch, will be worn to provide continuous physiological monitoring for safety. Participants will use the application by self-management for 9 months. All participants are given questionnaires, nutritional, physical fitness and physiological-biochemical assessment at baseline, 3 months, 6 months and 9 months.
  Arms: control group

SUMMARY:
Hypertension is a major risk factor for cardiovascular disease and cardiovascular events. Healthy lifestyle factors are widely recommended for hypertension prevention and control, and cardiorespiratory fitness is a strong and independent predictor of the progression of hypertension. Increased cardiorespiratory fitness through lifestyle modifications is associated with lower mortality in hypertensive or high-normal blood pressure individuals. The aim of the study is to evaluate the effects of supervised lifestyle intervention that include diet and exercise and base on intelligent application and continuous physiological monitoring on improvement of cardiopulmonary fitness, blood pressure and other health outcomes among participants with hypertension or high-normal blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. who is ≥18 years old and < 70 years old;
2. hypertension or high-normal blood pressure;
3. who has a smart phone and can use it (android phones are preferred).

Exclusion Criteria:

1. with acute myocardial infarction, acute tachyarrhythmia, pulmonary edema, severe aortic stenosis and other serious circulatory diseases or respiratory diseases;
2. with acute cardiovascular and cerebrovascular diseases;
3. poor blood pressure control;
4. with physical limitations(e.g., restricting injuries of the musculoskeletal system, such as fractures, unstable joints and other physical diseases);
5. with skin disease or skin damage at the site of wearable device;
6. with mental disorder, epilepsy or other diseases resulting in inability to control the body;
7. pacemaker installation;
8. woman who is during pregnancy or prepare for pregnancy;
9. sensitive skin for wearable devices; 10）refuse to provide written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-04-27 (Estimated); Study Completion 2023-10-27 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (VO2peak) from baseline to 3 months | baseline, 3 months
  VO2peak is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months.

SECONDARY OUTCOMES:
Change in systolic blood pressure | baseline, 3 months, 6 months and 9 months
  Systolic blood pressure is measured at baseline, 3 months, 6 months and 9 months. Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in diastolic blood pressure | baseline, 3 months, 6 months and 9 months
  Diastolic blood pressure is measured at baseline, 3 months, 6 months and 9 months. Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived anaerobic threshold (AT) | baseline, 3 months and 9 months
  AT is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived oxygen uptake efficiency slope (OUES) | baseline, 3 months and 9 months
  OUES is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived peak respiratory exchange ratio (RERpeak) | baseline, 3 months and 9 months
  RERpeak is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived VE/VCO2-slope | baseline, 3 months and 9 months
  VE/VCO2-slope is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived VO2/HR | baseline, 3 months and 9 months
  VO2/HR is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived total time of exercise | baseline, 3 months and 9 months
  Total time of exercise is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived peak metabolic equivalents (METs) | baseline, 3 months and 9 months
  Peak METs is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in cardiopulmonary exercise test-derived maximal heart rate | baseline, 3 months and 9 months
  Maximal heart rate is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in concentrations of serum lipids and lipoproteins | baseline, 3 months and 9 months
  Concentrations of serum lipids and lipoproteins, including low-density lipoprotein-cholesterol, total cholesterol, triglycerides, and high-density lipoprotein-cholesterol, are obtained from blood laboratory data, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in concentration of fasting serum glucose | baseline, 3 months and 9 months
  Concentration of fasting serum glucose is obtained from blood laboratory data, which is measured at baseline, 3 months and 9 months. Change from baseline to 3 months and 9 months will be measured.
Change in upper limb muscle endurance | baseline, 3 months, 6 months and 9 months
  The subject stands holding dumbbells (8 pounds for men, 5 pounds for women) with arms straight and hanging down next to the body. After the start, the subject will bend his arms to the shoulders and calculate 30 seconds. The total number of correct bends in 30 second. Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in lower limb muscle endurance | baseline, 3 months, 6 months and 9 months
  The subject sits in the middle of the chair with his back straight, hands crossed in front of his chest, after the start, the subject stands up and sits down, and counts the number of standing up and sitting times completed within 30 seconds. Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in handgrip strength | baseline, 3 months, 6 months and 9 months
  Adjust the grip bar so the second joint of the fingers fits snugly under the handle and takes the weight of the instrument. Set the dynamometer to zero. The subject holds the handgrip dynamometer in line with the forearm at the level of the thigh, away from the body. The subject squeezes the handgrip dynamometer as hard as possible without holding the breath. Neither the hand nor the handgrip dynamometer should touch the body or any other object. Repeat the test twice with each hand. The score is the highest of the two readings for each hand. Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in upper and lower limbs and body flexibility | baseline, 3 months, 6 months and 9 months
  The subject adopts a standing posture, with the dominant hand placed behind the shoulder on the same side, with the palm facing the back, with the fingers straight, stretch down as far as possible along the center of the back, and the palm of the other hand outwards from the bottom Extend your back upwards, keep your hands as close as possible, touch each other, or overlap your hands. Never hold and pull with your hands. Measure the distance between the middle finger of both hands.
  The subject sits on the front edge of the chair, with one foot bent on the ground, the other foot is straight forward, the heel touches the ground, the toes are raised, and the palms of both hands are folded (middle fingers) and stretched out. Stretch straight feet. Measure the distance from the middle finger to the toe.
  Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in balance ability | baseline, 3 months, 6 months and 9 months
  Stand with your hands on your waist, stand on one foot, and place the foot off the ground on the inside of the ankle that supports your foot. Record the right and left foot support time for correct actions, with a full score of 30 seconds.
  Change from baseline to 3 months, 6 months and 9 months will be measured.
Change in physical activity level | baseline, 3 months, 6 months and 9 months
  Average physical activity level is measured at baseline, 3 months, 6 months and 9 months by International Physical Activity Questionnaire (IPAQ). Daily physical activity level is recorded by worn smart watch. Change from baseline to 3 months, 6months and 9 months will be measured.
Change in dietary intake | baseline, 3 months, 6 months and 9 months
  Dietary intake is measured at baseline, 3 months, 6 months and 9 months by 24-hour dietary recalls for 3 days. Change from baseline to 3 months, 6months and 9 months will be measured.
Change in peak oxygen uptake (VO2peak) from baseline to 9 months | baseline, 9 months
  VO2peak is obtained by a graded cardiopulmonary exercise test to assess cardiorespiratory fitness, which is measured at baseline and 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Feng, MD PhD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No
to contact the researcher for sharing after the trial